CLINICAL TRIAL: NCT07120113
Title: Effect of Cupping Massage Versus Myofascial Release Therapy in Patients With Mechanical Neck Pain. A Randomized Controlled Trial
Brief Title: Effect of Cupping Massage Versus Myofascial Release Therapy in Patients With Mechanical Neck Pain
Acronym: neck pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Collaborators: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Sara Abdullah mohamed elsamahy, Lecturer of Physical Therapy, Misr University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MisrUniversity01
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2023-06

CONDITIONS: Mechanical Neck Pain
Keywords: mechanical neck pain
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cupping massage (Experimental): This group will receive cupping massage
  Interventions: Other: cupping massage
- myofascial release thechnique (Experimental): This group will receive myofascial release technique
  Interventions: Other: Myofascial release technique
- Control Group (Active Comparator): This group will receive traditional exercises
  Interventions: Other: Traditional exercises

INTERVENTIONS:
Other: cupping massage — This group will receive cupping massage three sessions per week for four weeks
  Arms: cupping massage
Other: Myofascial release technique — This group will receive the myofascial release technique three sessions per week for four weeks
  Arms: myofascial release thechnique
Other: Traditional exercises — This group will receive traditional exercises three sessions per week for four weeks
  Arms: Control Group

SUMMARY:
to investigate the effect of dynamic cupping versus myofascial release on pain level, range of motion and functional level in mechanical neck pain

ELIGIBILITY:
Inclusion Criteria:

* Body mass index less than or equal to 25kg/m2
* have had mechanical neck pain for at least the previous three months

Exclusion Criteria:

neck pain due to

* trauma
* disc propulsion
* congenital deformity
* spinal stenosis
* rheumatoid arthritis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
pain intensity | 0-3 month
  measuring by visual analog scale
Cervical Range of Motion | 0-1 month
  Cervical range of motion device

SECONDARY OUTCOMES:
functional level | 0-1 month
  Neck disability index measuring functional level

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt